CLINICAL TRIAL: NCT04113785
Title: In Vivo Kinematics for Subjects Implanted With Klassic TKA
Brief Title: In Vivo Kinematics for Subjects Implanted With Klassic Total Knee Arthroplasty (TKA)
Acronym: TKA
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Hofmann Arthritis Institute (Unknown); Duke University (Other)
Responsible Party: Principal Investigator, Richard Komistek, Principle Investigator, The University of Tennessee, Knoxville
Other Study IDs: WIRB20182087
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Total Knee Arthroplasty; Osteo Arthritis Knee; Knee Implant; Knee Injuries
Keywords: total knee arthroplasty; knee implant; osteoarthritis
MeSH Terms: conditions — Knee Injuries; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Klassic TKA: Subjects implanted with a Klassic TKA. Subjects will undergo flouoroscopic evaluation during a deep knee bend evaluation and the postoperative kinematics will be reported.
  Interventions: Device: Klassic Knee System

INTERVENTIONS:
Device: Klassic Knee System — At present, all TKA available for surgeons to use are asymmetric where there is a distinct femoral and tibial component for the left knee and a distinct femoral and tibial component for the right knee. The Klassic knee system is a symmetrical knee implant, where the same femoral and same tibial component can be used for either the right or left knee

SUMMARY:
In vivo knee kinematics will be assessed for 20 subjects that have been implanted with a Total Joint Orthopedics Klassic knee system by Dr. Aaron Hofmann of the Hofmann Arthritis Institute's Center for Precision Joint Replacement. This is the location from which all participants will be recruited and where fluoroscopy data collection will occur. Participants will undergo fluoroscopic surveillance of their implanted knee using a C-arm fluoroscopic unit while performing a deep knee bend activity at least six months post-operatively.

DETAILED DESCRIPTION:
Enrollment will be increased to 24 subjects to ensure that researchers acquire the necessary 20 usable datasets for analysis and also to account for any subjects that may drop out of the study. At present, all TKA available for surgeons to use are asymmetric where there is a distinct femoral and tibial component for the left knee and a distinct femoral and tibial component for the right knee. The Klassic knee system is a symmetrical knee implant, where the same femoral and same tibial component can be used for either the right or left knee. The kinematics for the 20 knees will be analyzed, including condylar roll-back, axial rotation, range of motion, and condylar lift-off

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will have a Klassic knee system.
2. Subjects must be at least six months post-operative.
3. Participants must be judged clinically successful with their most recent (new) Knee Society "Knee Score" equal to or greater than 80.
4. Participants must be able to perform a deep knee bend.
5. Subjects must be willing to sign the Informed Consent (IC) / HIPAA form to participate in the study.
6. Must speak English.

Exclusion Criteria:

1. Pregnant, potentially pregnant or lactating females. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study.
2. Subjects without the required type of knee implant.
3. Bilateral subjects (i.e., patients with both knees implanted)
4. Subjects who are unable to perform a deep knee bend.
5. Subjects who are unwilling to sign Informed Consent/ HIPAA documents.
6. Subjects who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Dr. Aaron Hofmann who have been implanted with the Klassic Knee System
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Komistek, Ph.D., Principal Investigator — The University of Tennessee
Locations (1):
- Hofmann Arthritis Institute for Precision Joint Replacement, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Researchers would like to retain this study data in our secure database so as to continue to add relevant, current data to our digital collection to help us work with manufacturers in the future to create better implants that last longer and will not require revision surgery. Participants will be asked if their study data may remain a part of the University of Tennessee's Center for Musculoskeletal Research data collection for use in future studies in the IC. Identifiers are automatically removed by the secure server after data are uploaded.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Klassic TKA
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Klassic TKA
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — The study did not collect age information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
  Between 18 and 65 years | NA — The study did not collect age information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
  >=65 years | NA — The study did not collect age information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — The study did not collect gender information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
  Male | NA — The study did not collect gender information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — The study did not collect race information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
  Asian | NA — The study did not collect race information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
  Native Hawaiian or Other Pacific Islander | NA — The study did not collect race information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
  Black or African American | NA — The study did not collect race information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
  White | NA — The study did not collect race information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
  More than one race | NA — The study did not collect race information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.
  Unknown or Not Reported | NA — The study did not collect race information as this was not of interest to the sponsor. Inclusion criteria included knee performance scores and postoperative time.

OUTCOME MEASURES:

1. Primary Outcome: Axial Rotation (AR) During Deep Knee Bend
Description: Rotation of femoral component with respect to tibial component during deep knee bend. Positive indicated external rotation of femur wrt tibia.
Time Frame: at least 6 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Klassic TKA
Number analyzed (Participants) | 21
degrees | 6.6 (3.2)

2. Primary Outcome: Maximum Weight-bearing Flexion During Deep Knee Bend
Description: Maximum weight-bearing flexion that the subjects are able to achieve during deep knee bend. All values are positive.
Time Frame: at least 6 months post-operative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Klassic TKA
Number analyzed (Participants) | 21
degrees | 111.7 (13.3)

3. Primary Outcome: Medial Condyle Translations During Deep Knee Bend Activity.
Description: Anterior Posterior (AP) translations of medial femoral condyle during deep knee bend. Positive indicates anterior sliding and negative indicates posterior rollback.
Time Frame: at least 6 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Klassic TKA
Number analyzed (Participants) | 21
mm | 2.5 (2.0)

4. Primary Outcome: Lateral Condyle Translations During Deep Knee Bend Activity
Description: Anterior Posterior (AP) translations of lateral femoral condyle during deep knee bend. Positive indicates anterior sliding and negative indicates posterior rollback.
Time Frame: at least 6 months post-operative
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Klassic TKA
Number analyzed (Participants) | 21
mm | 2.5 (2.0)

ADVERSE EVENTS:
Time Frame: at least 6 months post-operative
Arm/Group | Klassic TKA
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT04113785/Prot_SAP_000.pdf